CLINICAL TRIAL: NCT03483844
Title: Diagnostic Accuracy of Low-dose Dual-energy CT for the Pre-surgical Planning of Patients With Progression of Scoliosis
Brief Title: Low-dose Dual-energy CT for the Pre-surgical Planning of Patients With Progression of Scoliosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: TCbd17
Record Dates: First submitted 2018-03-07; First posted 2018-03-30 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Scoliosis
Keywords: scoliosis; low dose; arthrodesis; dual-energy CT
MeSH Terms: conditions — Scoliosis; Ankylosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: GE CT 750 HD — Low-dose dual-energy CT imaging

SUMMARY:
The aim of the study is to evaluate the diagnostic accuracy of low-dose dual energy CT in the pre-surgical planning of patients with progression of scoliosis

DETAILED DESCRIPTION:
CT imaging is the gold standard for assessing bone dysmorphism and vertebral morphometry during the pre-surgical planning of vertebral arthrodesis. It is necessary in the definition of the fixation points to avoid malposition of transpedicular screws and potential visceral, vascular or neurological damage.

It is known that multislice CT involves an increased radiation exposure for patients, while dual-energy CT uses a low-dose acquisition protocol and VEO reconstruction software.

The aim of the study is to evaluate the diagnostic accuracy of low-dose dual energy CT in the pre-surgical planning of patients with progression of scoliosis who are candidated for vertebral arthrodesis.

ELIGIBILITY:
Inclusion Criteria:

* patients with progression of scoliosis without vertebral arthrodesis
* patients able to maintain immobility for the duration of the exam
* patients from 5 to 20 years old

Exclusion Criteria:

* pregnancy
* vertebral arthrodesis
* patients unable to maintain immobility for the duration of the exam
* non-compliant patients
* obese patients
* patients younger than 5 years old or older than 20 years old

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with progression of scoliosis selected at the Rizzoli Orthopaedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Week 1 (post-surgery)
  To evaluate the percentage of malpositioning of transpedicular screw. A percentage of malpositioning lower than 10% will be considered as acceptable.

SECONDARY OUTCOMES:
Radiation exposure | Baseline (pre-surgery) and week 1 (post-surgery)
  Collection of dosimetric data

CONTACTS AND LOCATIONS:
Overall Officials: Milva Battaglia, MD, Principal Investigator — Rizzoli Orthopaedic Institute
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy